CLINICAL TRIAL: NCT02221232
Title: A Pilot Clinical Evaluation of the Antimicrobial Effectiveness of Topically Applied ZuraPrep™
Brief Title: Efficacy Study to Evaluate Antimicrobial Effectiveness of ZuraPrep™
Acronym: ZX-ZP-0035
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: To assess product performance (test and reference products), move into further testing.
Sponsor: Zurex Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 131112-103 (ZX-ZP-0035)
Record Dates: First submitted 2014-08-18; First posted 2014-08-20 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2014-11

CONDITIONS: Surgical Site Infection
Keywords: ZuraPrep; Antimicrobial; Bio-Science Laboratories; Zurex Pharma; Surgical/Patient preoperative skin preparation
MeSH Terms: conditions — Surgical Wound Infection | interventions — chlorhexidine gluconate; 2-Propanol; Chromogranins; citrate, isopropyl alcohol, methylene blue, parabens drug combination; Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- ZuraPrep Config 1 (Experimental): Isopropyl alcohol (IPA) 70% Standard scrub time.
  Interventions: Drug: ZuraPrep
- ZuraPrep Config 2 (Experimental): Isopropyl alcohol (IPA) 70% Half scrub time.
  Interventions: Drug: ZuraPrep
- ZuraPrep Vehicle (Placebo Comparator): ZuraPrep without IPA
  Interventions: Drug: ZuraPrep Vehicle
- ChloraPrep (Active Comparator): Chlorhexidine gluconate (CHG) 2% / Isopropyl alcohol (IPA) 70%
  Interventions: Drug: Chloraprep

INTERVENTIONS:
Drug: Chloraprep — Apply topically.
  Other Names: 2% chlorhexidine gluconate / 70% Isopropyl alcohol; CHG 2% / IPA 70%
  Arms: ChloraPrep
Drug: ZuraPrep — Apply topically.
  Other Names: Isopropyl alcohol 70%
  Arms: ZuraPrep Config 1; ZuraPrep Config 2
Drug: ZuraPrep Vehicle — Apply topically.
  Other Names: ZuraPrep without IPA; ZuraPrep Placebo
  Arms: ZuraPrep Vehicle

SUMMARY:
The purpose of this pilot study is to evaluate antimicrobial properties of a single test product, a vehicle product and a reference product applied in two different areas when used as a patient preoperative skin preparation.

DETAILED DESCRIPTION:
This is an open label pilot study to evaluate antimicrobial properties of a single test product, a vehicle product and a reference product applied bilaterally to the skin of the abdomen and the inguina. Testing will be performed according to FDA TFM for Effectiveness Testing of a Patient Preoperative Skin Preparation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects may be of either sex, at least 18 years of age and of any race.
* Subjects must be in good general health, as evidenced by the Subject Confidential Information and Acceptance Criteria
* Subjects must read and sign an Informed Consent Form, Authorization to Use and Disclose Protected Health Information Form, and List of Restricted Products

Exclusion Criteria:

* Exposure of test sites to antimicrobial agents, medicated soaps, medicated shampoos, or medicated lotions, use of biocide-treated pools or hot tubs, use of tanning beds, or sunbathing during the 14-day pre-test conditioning period or during the test period.
* Use of topical or systemic antimicrobials, antibiotics, or steroids (other than hormones for contraception or post-menopausal indications), or any other product known to affect the normal microbial flora of the skin during the 14-day pre-test conditioning period or during the test period.
* Exposure of the test sites to strong detergents, solvents, or other irritants during the 14-day pre-test conditioning period or during the test period.
* Known allergies to vinyl, latex (rubber), alcohols, metals, inks, or tape adhesives, or to common antibacterial agents found in soaps, lotions, or ointments, particularly chlorhexidine gluconate (CHG), citric acid, methylene blue, methylparaben, propylparaben, or isopropyl alcohol.
* A medical diagnosis of a physical condition, such as a current or recent severe illness, asthma, diabetes, hepatitis, an organ transplant, mitral valve prolapse, congenital heart disease, internal prostheses, or any immunocompromised conditions such as AIDS (or HIV positive).
* Subjects must be unable to become pregnant, or willing to use an acceptable method of contraception to prevent pregnancy, if female of child-bearing potential.

Inability to become pregnant would include subjects who are:

* Male
* Females unable to become pregnant (i.e., postmenopausal for at least 1 year or surgically sterile due to hysterectomy, bilateral oophorectomy, uterine ablation, or bilateral tubal ligation)
* Females of child-bearing potential but using acceptable methods of contraception, including one of the following methods that have been used for at least 2 weeks prior to Treatment Day Visit.

Acceptable methods of contraception include one of the following methods:

* Systemic birth control (the same type of birth control for at least 3 months prior to entering the study and continuation of this type of birth control throughout the study)
* Double barrier methods (condom with spermicide or diaphragm with spermicide)
* IUD
* Vasectomized partner; or
* Abstinence from sexual intercourse

  * Any large tattoos, scars, active skin rashes, or breaks in the skin of the test sites.
  * Dermatoses, cuts, lesions, or other skin disorders on or around the test sites
  * A currently active skin disease or inflammatory skin condition (e.g., contact dermatitis) that, in the opinion of the Consulting Physician or Principal Investigator, would compromise subject safety or study integrity.
  * Showering, bathing, or swimming within the 72 hour period prior to Baseline Day, the first Test Day, and throughout the test period.
  * Participation in another clinical study in the past 30 days or current participation in another clinical study.
  * Any medical condition or use of any medications that, in the opinion of the Medical Expert/Consulting Physician or Principal Investigator, should preclude participation.
  * Unwillingness to fulfill the performance requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Calculations of mean log10 reductions from baseline populations | 0-24 hours post dose
  Antimicrobial efficacy will be evaluated based upon calculation of mean log10 reductions from baseline populations by subtracting the log10 number of viable microorganisms recovered at each post-product application sample from the log10 number of viable microorganisms recovered in the baseline samples. The performance criteria are mean reductions in microbial flora of ≥2 log10 per square cm on skin of the abdomen and ≥3 log10 per square cm on skin of the inguen.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Beausoleil, Principal Investigator — BioScience Laboratories, Inc.
Locations (1):
- BioSciences Laboratories, Inc., Bozeman, Montana, United States